CLINICAL TRIAL: NCT00543478
Title: Role Of Saccharomyces Boulardii In Diarrhea Dominant Irritable Bowel Syndrome
Brief Title: Saccharomyces Boulardii in Diarrhea Dominant Irritable Bowel Syndrome
Acronym: SBIBS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aga Khan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SB; URC 071006MED
Record Dates: First submitted 2007-10-12; First posted 2007-10-15 (Estimated); Last update posted 2007-10-15 (Estimated); Status verified 2007-10

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable bowel syndrome; Diarrhea; Probiotics
MeSH Terms: conditions — Irritable Bowel Syndrome; Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Receive active drug Saccharomyces boulardii 250mg twice a day for 8 weeks.
  Interventions: Drug: Saccharomyces boulardii
- 2 (Placebo Comparator): Placebo will be given twice a day for 10 weeks
  Interventions: Drug: Methyl cellulose powder (low viscosity)

INTERVENTIONS:
Drug: Saccharomyces boulardii — 250mg, twice a day in sachets, for 8 weeks
  Arms: 1
Drug: Methyl cellulose powder (low viscosity) — twice a day sachets for 10 weeks
  Arms: 2

SUMMARY:
Probiotics are friendly bacteria normally present in food products like yogurt whereas irritable bowel syndrome is a longstanding functional disorder characterized by abdominal pain and altered bowel habits either diarrhea or constipation dominant without a definitive etiology.

Study Hypothesis:Does probiotics(Saccharomyces boulardii improves daily bowel symptoms and quality of life in patients with diarrhea dominant irritable bowel syndrome?

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is a common functional disorder and may lead to impaired social and personal function and can diminish quality of life.While the precise pathophysiology of IBS remains to be elucidated, dysmotility and altered visceral sensory perception are currently the most popular hypothesis. There has been a suggestion that some patients with IBS may harbor bacterial overgrowth leading to low grade inflammation, immune activation, and their symptoms may be ameliorated by its eradication.Probiotics, defined as live or attenuated bacteria or micro organism that confer a significant health benefit to the host.

* I. Firstly, probiotic organism exert antibacterial and antiviral effects.
* II. Probiotics could alter the composition of the gut flora, either directly through augmentation of commensal or indirectly through a reduction in pathogen related inflammation or bacterial fermentation.

Trial protocol:

Phase 1: placebo BID (1 week),both arms Phase 2: Randomization by pharmacy, placebo vs. active drug (6 weeks) Phase 3: placebo BID (1 week), both arms

-III. Probiotics have been demonstrated to exert anti-inflammatory effects at mucosal surfaces by reducing mucosal inflammation, decreasing immune mediated activation of enteric motor and sensory neurons and modifying neural traffic between the gut and central nervous system.

Saccharomyces Boulardii is a probiotic yeast and its role for the treatment of IBS has not been extensively investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be recruited from gastroenterology clinic at Aga Khan University hospital with diagnosis of diarrhea dominant irritable syndrome.
* Age between 18- 60 years.
* Male and female both.
* Organic gastrointestinal diseases excluded by baseline laboratory and sigmoidoscopy/colonoscopy and biopsy within last 2 years.
* All Patients need to satisfy ROME III criteria

Exclusion Criteria:

* Age < 18 and > 60 years
* Pregnant and lactating females
* Patients on laxatives or antidiarrheal drugs that could influence the motility of gut
* Patient on antibiotics or within 2 weeks of starting protocol.
* Not willing to participate
* Non-compliant in run in period.
* Patients taking Husk.
* Diabetic patients

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2007-10; Study Completion 2008-07 (Estimated)

PRIMARY OUTCOMES:
Any Improvement in symptoms of number of bowel habits, urgency, straining,sense of incomplete evacuation, stool form (evaluated by Bristol stool form scale, abdominal pain and bloating/flatulence | 10 weeks

SECONDARY OUTCOMES:
Improvement in quality of life in diarrhea dominant IBS by validated IBS-QOL questionnaire. | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lubna Kamani, FCPS,MRCP, Principal Investigator — Aga Khan University
Locations (1):
- Gastroenterology outpatients clinics,Aga Khan University hospital, Karachi, Pakistan